CLINICAL TRIAL: NCT02859090
Title: Single-centre Study of the Expression of Heat Shock Proteins in the Lymphocytes From the Tonsils of Patients With Various Diseases Requiring Tonsillectomy
Brief Title: Study of the Expression of Heat Shock Proteins in Populations of B Lymphocytes in Human Tonsils
Acronym: HOTLYMPHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: DUVILLARD UB 2012
Record Dates: First submitted 2016-08-04; First posted 2016-08-08 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Tonsillectomy
MeSH Terms: interventions — Tonsillectomy; Blood Specimen Collection

ARMS (1):
- patient (Experimental)
  Interventions: Procedure: tonsillectomy; Biological: blood sample

INTERVENTIONS:
Procedure: tonsillectomy
Biological: blood sample

SUMMARY:
It has recently been shown that various HSPs are strongly expressed in B lymphomas. Indeed, HSP90 stabilizes the protein Bcl-6 in diffuse large-cell B lymphomas. Pharmacological inhibition of HSP90 in vitro induced apoptosis in lymphoma cells (Cerchietti et al. Nat. Medicine, 2009, 1369-1376). In addition, HSP110 is strongly expressed in non-Hodgkin lymphomas, and targeting this HSP at the cell surface using specific antibodies could constitute a future therapy (Zappasodi et al. Blood, 2011, 4421-4430). Despite the importance of these proteins in the development of lymphomas, their expression and their role in the activation of normal B lymphocytes and the normal development of germinal centres is not known.

The expression of Heat shock proteins should vary among the different B lymphocyte populations present in the tonsils (naïve B cells, memory B cells, germinal centre B cells).

The aim of this study is to establish an expression profile for heat shock proteins in populations of B lymphocytes in human tonsils

ELIGIBILITY:
Inclusion Criteria:

* Persons who have provided oral consent
* Tonsillectomy in children or adults

Exclusion Criteria:

* Persons without national health insurance cover
* Adults under guardianship
* Pregnant or breast-feeding women
* Persons with positive HIV or HCV serology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-08-26 (Actual); Primary Completion 2014-11-20 (Actual); Study Completion 2014-11-20 (Actual)

PRIMARY OUTCOMES:
expression of heat shock proteins | Day one

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France